CLINICAL TRIAL: NCT01278485
Title: Naturalistic Evaluation of Hypoglycemic Events in Diabetic Subjects
Brief Title: Evaluation of Low Blood Sugar Events in Participants With Diabetes (MK-0431-402)
Acronym: NEEDS
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-402
Record Dates: First submitted 2011-01-13; First posted 2011-01-19 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sulphonylurea (SU) Monotherapy or SU + Metformin: Participants with Type 2 diabetes that have been treated with SU monotherapy for at least 6 months by a cardiologist, nephrologist, or family practice doctor.
  Interventions: Drug: Sulphonylurea; Drug: Metformn

INTERVENTIONS:
Drug: Sulphonylurea — SU administered according to usual practice.
Drug: Metformn — Metformin administered according to usual practice.

SUMMARY:
This is a multicenter, observational, retrospective and cross-sectional study to be conducted in a cohort of consecutively selected participants with type 2 diabetes mellitus (T2DM) who have been treated with sulphonylurea (SU) monotherapy or SU + metformin (MF) combination therapy by their cardiologist, nephrologist, or family practice doctor for at least 6 months prior to study enrollment.

The purpose of the study is to assess treatment patterns, goal attainment rates, long-term diabetes complication rates, and frequency and severity of hypoglycemic episodes among T2DM participants treated in cardiology, nephrology and family practice settings.

ELIGIBILITY:
Inclusion Criteria

* Participants diagnosed with type 2 diabetes mellitus (DM).
* Participants at least 30 years of age at time of type 2 DM diagnosis.
* Participants treated with SU monotherapy or SU + MF combination therapy for at least 6 months prior to enrollment.
* Participants receiving diabetes care from a cardiologist, nephrologist or family practitioner for at least 6 months.
* Participants with a clinical record in the health care center.
* Participants in whose medical records a minimum core data set can be found; core data defined as: age, gender, duration of diabetes/age at diagnosis, all glucose-lowering medications (branded and generic names, dosage, dosing frequency, starting and stopping dates) since the start of all antihyperglycemic medications.

Exclusion Criteria

* Participants with Type 1 DM.
* Participants who are pregnant or with gestational DM.
* Participants receiving any anti-diabetic treatment from an endocrinologist/diabetologist in the previous 6 months.
* Participants requiring daily concomitant usage of insulin.
* Participants receiving any other oral diabetes medications other than SU or SU + MF.
* Participants who are already participating in a clinical trial or other clinical study.
* Participants for whom it would be impossible to complete the questionnaire.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Type 2 diabetes mellitus ≥30 years of age who have been treated with sulphonylurea (SU) monotherapy or SU+ merformin (MF) combination therapy for at least 6 months by a cardiologist, nephrologist, or family practice doctor.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled a total of 726 Korean participants who had been treated with sulfonylurea monotherapy or sulfonylurea and metformin combination therapy for at least six months in the departments of Cardiology, Nephrology, and Family Medicine of various Korean hospitals and medical centers.
Pre-assignment Details: Seven participants who failed to meet all the inclusion criteria were excluded from the study.
Groups:
- Adults With Type 2 Diabetes Mellitus ≥30 Years of Age: Adults with Type 2 diabetes mellitus ≥30 years of age who have been treated with sulphonylurea (SU) monotherapy or SU+ metformin (MF) combination therapy for at least 6 months by a cardiologist, nephrologist, or family practice doctor.
Period: Overall Study
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Started | 719
Completed | 719
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 719
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.91 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319
  Male | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Hypoglycemic Episodes in the 6 Months Prior to Enrollment
Description: The participant experience of low blood sugar (hypoglycemia) questionnaire was used to evaluate participants' experience of hypoglycemia during the previous 6 months. Participants were asked to record whether they experienced hypoglycemia symptoms (yes/no) and to record the severity of those symptoms as mild, moderate, severe, or very severe.
Time Frame: Up to 6 Months Prior to Enrollment
Population: All enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 719
Participants | 305

2. Primary Outcome: Number of Participants Experiencing Mild, Moderate, Severe, or Very Severe Hypoglycemic Episodes in the 6 Months Prior to Enrollment
Description: At the time of enrollment, participants were asked to rate their hypoglycemic episodes in the last 6 months as mild, moderate, severe, or very severe. Participants were able to select more than one category.
Time Frame: Up to 6 Months Prior to Enrollment
Population: All enrolled participants that experienced hypoglycemia in the prior 6 months.
Measure: Number; unit: Participants
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 305
Participants
  Mild | 279
  Moderate | 93
  Severe | 91
  Very Severe | 28

3. Secondary Outcome: Participant Mean Score on the EuroQol-5 Dimension (EQ-5D) Quality-of-Life Questionnaire At the Time of Enrollment
Description: The EQ-5D is a questionnaire that assesses participant quality of life in 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has 3 levels: no problems, some problems, extreme problems for which participants are asked to self-rate their experience. The EQ-5D total score ranges from -0.171 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
Time Frame: Day of Enrollment
Population: All enrolled participants with a completed EQ-5D questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 714
Score on a Scale | 0.89 (0.14)

4. Secondary Outcome: Participant Mean Score on the EuroQol Visual Analog Scale (EQ-VAS) Quality-of-Life Questionnaire At the Time of Enrollment
Description: Participant health status was self-reported in 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and was analyzed by using visual analog scale (VAS) which records participant responses on a scale of 0 (poor health) to 100 (excellent health).
Time Frame: Day of Enrollment
Population: All enrolled participants with a completed EQ-VAS questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 714
Score on a Scale | 72.10 (16.68)

5. Secondary Outcome: Participant Mean Score on the Treatment Satisfaction Questionnaire for Medication (TSQM) At the Time of Enrollment
Description: The TSQM is a treatment satisfaction questionnaire containing 14 items covering the following dimensions: side effects, effectiveness, convenience, and global satisfaction. Participants were asked to respond in a yes or no fashion, or by using a 5- or 7-point Likert scale. The score for each dimension ranges from 0 to 100, with a higher score expressing a better quality of life.
Time Frame: Day of Enrollment
Population: All enrolled participants that completed the TSQM on the day of enrollment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 716
Score on a Scale
  Effectiveness | 64.48 (12.96)
  Side Effects | 97.18 (10.63)
  Convenience | 67.71 (13.38)
  Global Satisfaction | 63.08 (14.46)

6. Secondary Outcome: Participant Mean Score on the Self-Reported Adherence and Barriers Questionnaire At the Time of Enrollment
Description: The self-reported adherence and barriers questionnaire to measure treatment compliance asked participants to rate their responses to 5 questions: How often do you take your diabetes medicines exactly as your healthcare provider prescribes them?; During the past 4 weeks, how often were you unsure about some of the things your doctor suggested you do for your diabetes?; During the past 4 weeks, how often were you unable to do what was necessary to follow your doctor's treatment plans for your diabetes?; During the past 4 weeks, how often were you bothered by side effects from your medicines?; and During the past 4 weeks, how often did you have problems getting your prescriptions filled? Participants responded using a scale of 1 to 5, where 1=always, 2=usually, 3=sometimes, 4=rarely, and 5=never.
Time Frame: Day of Enrollment
Population: All enrolled participants that completed a questionnaire on the day of enrollment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 719
Score on a Scale
  Takes Medicine Exactly As Prescribed (n=719) | 1.54 (0.81)
  Unsure About Treatment Plan Last 4 Weeks (n=719) | 4.32 (1.10)
  Followed Treatment Plan Last 4 Weeks (n=718) | 3.95 (1.14)
  Problems With Side Effects Last 4 Weeks (n=711) | 4.85 (0.53)
  Problem Filling Prescriptions Last 4 Weeks (n=719) | 4.92 (0.43)

7. Primary Outcome: Number of Participants With Hemoglobin A1c <7.0% at the Time of Enrollment
Description: Participant serum samples were collected after an overnight fast to determine the hemoglobin A1c level. Hemoglobin A1c is a measure of the percentage of glycated hemoglobin in the blood and provides an indication of participant blood glucose control in the 2 to 3 months prior to the evaluation.
Time Frame: Day of Enrollment
Population: All enrolled participants with a hemoglobin A1c measurement collected on the day of enrollment.
Measure: Number; unit: Participants
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 717
Participants | 404

8. Secondary Outcome: Participant Mean Score on the Worry Scale of Hypoglycemia Fear Survey (HFS II) At the Time of Enrollment
Description: Fear about hypoglycemia during 6 months prior to enrollment was evaluated using the Worry Scale of the HFS II. Responses to the 18-item questionnaire were recorded on a 0 to 4 scale, with 0=never, 1=rarely, 2=sometimes, 3=often, 4=almost always. The total score ranges from 0 to 72, with higher scores indicating increasing fear of hypoglycemia.
Time Frame: Day of Enrollment
Population: All enrolled participants that completed the worry scale of the HFS II.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 709
Score on a Scale | 6.98 (11.27)

9. Secondary Outcome: Number of Participants Experiencing a Change in Body Weight in the 12 Months Prior to Enrollment
Description: Participants were asked to rate their weight change experience in the 12 months prior to enrollment as: weight increased, weight decreased, or weight remained stable.
Time Frame: Up to 12 Months Prior to Enrollment
Population: All enrolled participants
Measure: Number; unit: Participants
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 719
Participants
  Gained Weight | 115
  Lost Weight | 148
  Weight Remained Stable | 456

10. Secondary Outcome: Number of Participants Reporting Body Weight Fears in the 12 Months Prior to Enrollment
Description: On the day of enrollment, participants were asked to rate their fear of gaining weight in the 12 months prior to enrollment using a self-administered questionnaire. The questionnaire elicited responses to 3 statements (I worry about gaining weight; I worry that my diabetic treatment makes me gain weight; and I worry about not being able to stabilize my weight) and relied on a scale of 0 to 4, where 0=never, 1=rarely, 2=sometimes, 3=often, and 4=almost always.
Time Frame: Up to 12 Months Prior to Enrollment
Population: All enrolled participants that completed the fear of weight gain questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Number analyzed (Participants) | 716
Score on a Scale
  Worries About Gaining Weight | 1.18 (1.36)
  Worries Diabetic Treatment Causes Weight Gain | 0.93 (1.26)
  Worries About Inability to Stabilize Weight | 0.93 (1.26)

ADVERSE EVENTS:
Description: Adverse event reporting was not planned nor evaluated for participants.
Arm/Group | Adults With Type 2 Diabetes Mellitus ≥30 Years of Age
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No